CLINICAL TRIAL: NCT01523600
Title: Effect of Whole Body Vibration Training on Physical Functioning and Risk of Falling in Older People Using Sheltered Housing
Brief Title: Whole Body Vibration Training Among Older People Using Sheltered Housing
Acronym: VAREX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: UKK Institute (Other)
Collaborators: Ministry of Education and Culture, Finland (Other); Pirkanmaa Hospital District (Unknown)
Responsible Party: Principal Investigator, Harri Sievanen, Research Director, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 138,04; R11122 (Other: Ethics Committee)
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Falls; Physical Performance; Fear of Falling
Keywords: whole body vibration; physical functioning; falls; older people; prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole body vibration training (Experimental)
  Interventions: Behavioral: Whole body vibration training
- Wellness group (Active Comparator)
  Interventions: Behavioral: Wellness group

INTERVENTIONS:
Behavioral: Whole body vibration training — The intervention comprises a 10-week individually supervised, progressive WBV training done twice a week on a side-alternating device with simultaneous body transferring and slight squatting exercises. At the week one, the duration of a single training bout is 1 x 1 min, and the number of 1 min bouts is weekly increased by one until five bouts is reached. During weeks 4 - 10, the training comprises 5 x 1 min bouts with 1 min rest periods between. During weeks 1 to 3, vibration frequencies are 12 and 18 Hz, which are used alternately. Thereafter, also 26 Hz may be used instead of 18 Hz. In addition, the amplitude of vibration is increased progressively according to a specified protocol. A detailed training diary is kept.
  Other Names: Galileo Med M Plus
  Arms: Whole body vibration training
Behavioral: Wellness group — The intervention comprises a 10-week supervised group training done once a week with the focus on stretching and flexibility exercises done mostly in a sitting position. The duration of a single training session is 45 minutes. A training diary is kept.
  Arms: Wellness group

SUMMARY:
The purpose of this randomised (double-blind) controlled exercise intervention trial is to determine whether the whole body vibration (WBV) training can effectively improve physical functioning of older people living in or regularly using services of sheltered housing, reduce their fear of falling, and prevent falling. The study comprises a 10-week training period and a 10-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* lives in sheltered housing or uses regularly services provided by sheltered housing
* ambulatory, able to walk independently with or without a walking aid
* Mini Mental State Examination (MSSE) points 16 or more

Exclusion Criteria:

* knee or hip prosthesis
* osteosynthetic material in lower limbs
* stiffening operation of the spinal column
* cardiac pacemaker
* recent fracture (< 1 yr for lower limb or spinal fractures, < ½ yr for upper limb fractures)
* recent major surgical operation
* acute thrombosis or its high risk
* acute musculoskeletal inflammation
* gall or bladder stones
* problematic hernia
* unstable cardiovascular or other systematic disease
* tumor
* diabetic neuropathy
* strong vertigo

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of falls | One year
  Participants keep fall diaries on daily basis and mail the diaries to the investigators in every month. In case of a reported fall, the investigator contacts the participant and enquires the details of the fall.

SECONDARY OUTCOMES:
Physical functioning | 10 weeks and one year
  The standard Short Physical Performance Battery (SPPB) is used for the assessment of participant's balance, walking speed and chair rising time at the baseline, after the 10 week training and after the subsequent 10 month follow-up.In addition, 4-m maximal walking speed , Timed Up and Go (TUG) test and grip strength are assessed at the same time points.
Fear of falling | 10 weeks and one year
  The Falls Efficacy Scale (FES-I)is used for the assessment of perceived fear of falling at the baseline, after 10 week training and after the subsequent 10-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Harri Sievanen, ScD, Study Director — The UKK Institute
Locations (4):
- Finland (4):
  - Kaukaharjun Seniorikeskus, Tampere
  - Kuuselan Seniorikeskus, Tampere
  - Tammenlehvä-keskus, Tampere
  - Viola-koti, Tampere